CLINICAL TRIAL: NCT00855088
Title: A Phase IV, Open Label Study in Healthy Male Subjects to Investigate the Extent of Darunavir/Ritonavir and Etravirine Exposure in Blood, Seminal Fluid, and Rectal Mucosal Tissue Following Single and Multiple Dosing of Darunavir/Ritonavir and Etravirine
Brief Title: Study in Healthy Males to Measure Darunavir and Etravirine in Blood, Seminal Fluid, and Rectal Tissue
Acronym: DESeRT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Tibotec Pharmaceutical Limited (Industry)
Responsible Party: Angela Kashuba, PharmD, UNC Chapel Hill Eshelman School of Pharmacy
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UNC IRB 08-0419
Record Dates: First submitted 2009-03-02; First posted 2009-03-04 (Estimated); Last update posted 2011-05-13 (Estimated); Status verified 2011-05

CONDITIONS: HIV/AIDS; HIV Infections
Keywords: HIV seronegativity
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections | interventions — Darunavir; Ritonavir; etravirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Darunavir, ritonavir, etravirine (Experimental): Single arm trial looking at the pharmacokinetics of darunavir, ritonavir, etravirine in healthy volunteers.
  Interventions: Drug: darunavir; Drug: Ritonavir; Drug: Etravirine

INTERVENTIONS:
Drug: darunavir — Healthy male volunteers will take darunavir 600 mg orally twice daily for 15 doses (8 days)
  Other Names: Prezista
Drug: Ritonavir — Healthy male volunteers will take ritonavir 100 mg orally twice daily for 15 doses (8 days)
  Other Names: Norvir
Drug: Etravirine — Healthy male volunteers will take etravirine 200 mg orally twice daily for 15 doses (8 days)
  Other Names: Intelence

SUMMARY:
This study is being conducted to look at how the body handles the drugs darunavir and etravirine. It will measure the amount of darunavir and etravirine in blood, semen, and in the rectum of men. The aim is to understand how much of the drug (taken by mouth) reaches the reproductive and intestinal tracts. It is believed that the presence of this drug in these areas may be beneficial in preventing the AIDS virus (HIV) from being passed from one person to another. The study will take samples of blood, semen and rectal mucosal tissue to measure drug levels. This study will also collect information on side effects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between the ages of 18 and 49 years, inclusive, with intact genital tract and gastrointestinal tract. (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG for individuals >35yo and clinical laboratory tests).
* Body Mass Index (BMI) of approximately 18 to 30 kg/m2; and a total body weight >/=50 kg (110 lbs).
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the trial.
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Subjects with a history of having a gastrectomy, colostomy, ileostomy, or any other procedure altering the gastrointestinal tract.
* Subjects with inflammatory bowel diseases (ulcerative colitis or Crohn's disease) and have a clearly defined diagnosis of irritable bowel syndrome.
* Subject who is unwilling to refrain from any sexual activity including intercourse and masturbation for 72 hours prior study visit Day 1 and until discharge from the study.
* Subject who is unwilling to refrain from rectal insertion of medical/recreation devices and products and from receptive anal intercourse, for 72 hours before study visit Day -1 and through 7 days after the last biopsy unless instructed otherwise by the investigators.
* History of febrile illness within 5 days prior to the first dose.
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug screen.
* A positive result for HIV.
* Active hepatitis B infection as defined by a positive Hepatitis B surface antigen (HbsAg) OR a positive Hepatitis B core antibody with a negative Hepatitis B surface antibody (HBsAb).
* Active hepatitis C infection as defined by anti-hepatitis C virus serology (as determined by multi-antigen EIA) and detectable HCV RNA.
* A positive test for syphilis, gonorrhea, Chlamydia, HSV-2 (active lesions) or trichomonas at screening.
* History of regular alcohol consumption exceeding 14 drinks (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of spirits) per week.
* Participation in a clinical study within 4 months preceding the first dose of trial medication.
* Participation in a rectal biopsy study in the 12 months preceding the first dose of trial medication.
* Use of prescription or nonprescription drugs, vitamins and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of trial medication. Herbal supplements must be discontinued 14 days prior to the first dose of trial medication. As an exception, acetaminophen may be used at doses of </= 1 g/day
* Blood donation of approximately 1 pint (500 mL) within 56 days prior to dosing.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Unwilling to abstain from alcohol use from 24 hours prior to the first dose of study medication until after the follow-up visit.
* Unwilling to abstain from cigarette smoking completely during inpatient pharmacokinetic visits and unwilling to limit smoking to a maximum of 5 cigarettes per day from 24 hours prior to the start of the study until study completion.
* Unwilling or unable to comply with the dietary restrictions in regard to study drug administration

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2009-07; Primary Completion 2010-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
To generate individual pharmacokinetic parameters for darunavir, ritonavir, and etravirine in seminal plasma after single and multiple dosing | Study days 1, 7, and 8
To generate composite pharmacokinetic parameters for darunavir, ritonavir, and etravirine in rectal tissue after single and multiple dosing | Study days 1 and 7 or 8

SECONDARY OUTCOMES:
To generate matrix:blood plasma ratios of darunavir, ritonavir, and etravirine in semen and rectal tissue after single and multiple dosing | Study days 1, 7 and 8

CONTACTS AND LOCATIONS:
Overall Officials: Angela DM Kashuba, PharmD, Principal Investigator — UNC Eshelman School of Pharmacy; Kristine B Patterson, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Hospitals CTRC, Chapel Hill, North Carolina, United States